CLINICAL TRIAL: NCT03184480
Title: Arnuity Ellipta Drug Use Investigation
Brief Title: Arnuity® Ellipta® Drug Use Investigation
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 207580
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Asthma
Keywords: Drug Use Investigation; GW685698; asthma; Post-marketing surveillance; ARNUITY ELLIPTA
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SUBJECTS RECEIVING ARNUITY ELLIPTA: Subjects with a diagnosis of asthma bronchial, for which Arnuity is indicated, who are naïve to Arnuity will be included.
  Interventions: Drug: Arnuity Ellipta

INTERVENTIONS:
Drug: Arnuity Ellipta — The active component of Arnuity Ellipta is fluticasone furoate and it is indicated for the treatment of bronchial asthma. Post-marketing investigation of ARNUITY ELLIPTA will be carried out in this analysis.

SUMMARY:
The aim of this post-marketing investigation is to collect and assess the information about safety and effectiveness of ARNUITY® ELLIPTA® (hereinafter referred to as "Arnuity") in daily clinical practice. The investigation will include subjects with a diagnosis of asthma bronchial who are naïve to ARNUITY. The investigator will monitor the information about safety and effectiveness of ARNUITY for one year from the start date of ARNUITY administration and Pneumonia will be considered as the priority investigation matter. 300 subjects, from approximately 150 medical institutions, will be included in this analysis. ARNUITY ELLIPTA is the registered trademark of GlaxoSmithKline (GSK) group of companies.

ELIGIBILITY:
Inclusion Criteria:

* The investigation will include subjects with a diagnosis of asthma bronchial, for which Arnuity is indicated and who are naïve to Arnuity.

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigation will assess the information about safety and effectiveness of Arnuity in approximately 300 subjects with a diagnosis of asthma bronchial, for which Arnuity is indicated and who are naïve to Arnuity.
Sampling Method: Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2017-08-19 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs), serious AEs (SAEs), severe AEs and drug related AEs | One year from the start of Arnuity administration
  The investigator will collect the information about all AEs (e.g., a disease, symptom, abnormal laboratory value) occurring after the start of Arnuity administration, regardless of whether or not Arnuity is related to an AE.
Number of subjects with pneumonia | One year from the start of Arnuity administration
  Pneumonia will be considered as priority investigation matter for this investigation and its occurrence will be monitored throughout the study period.
Response rate based on global assessment of effectiveness | One year from the start of Arnuity administration
  The response rate is the proportion of subjects assessed as "effective". Effectiveness will be comprehensively assessed based on the course of subjective and clinical symptoms and changes in Asthma Control Test (ACT) scores, etc. from the start date of administration to the end of the observation period.
Total ACT score | One year from the start of Arnuity administration
  ACT is a simple 5-question tool to evaluate the progression of asthma. Investigator will record the information from the ACT completed by subjects at the start of Arnuity administration, at Month 3, Year 1 from the start of Arnuity administration, or at the time of withdrawal from/termination of administration.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Nagasaki